CLINICAL TRIAL: NCT03314558
Title: Has Pulmonary Rehabilitation a Positive Impact on Sleep Quality in Patients Suffering From Chronic Obstructive Pulmonary Disease?
Brief Title: Has Pulmonary Rehabilitation a Positive Impact on Sleep Quality in Patients Suffering From COPD ?
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, Chef de Clinique, Centre Hospitalier Universitaire Saint Pierre
Other Study IDs: RR2017
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: COPD
Keywords: COPD; pulmonary rehabilitation; insomnia; sleep quality; physical activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients following a pulmonary rehabilitation program: COPD patients following a pulmonary rehabilitation program
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Other: pulmonary rehabilitation — a pulmonary rehabilitation program of 30 sessions, (3X1h/ week), will be followed by the COPD patients

SUMMARY:
The purpose of our study is to assess the impact of pulmonary rehabilitation on objective sleep quality in COPD patients.

DETAILED DESCRIPTION:
COPD patients suffer from bad sleep quality. About 27 -50% are suffering from insomnia, and respiratory related symptoms are also inducing sleep disturbances. Recently, a correlation between altered sleep quality and low activity levels have been shown in this population. In primary insomnia, it is well established that physical activity has a positive impact on sleep quality.

The purpose of our study is to assess the impact of pulmonary rehabilitation on objective sleep quality in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients
* able to walk and cycle

Exclusion Criteria:

* Shift work
* orthopedic diseases of limbs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients physically able to follow a pulmonary rehabilitation program
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
sleep efficiency | 3 +/- 2 months
  sleep efficiency assessed by actigraphy

SECONDARY OUTCOMES:
steps | 3 +/- 2 months
  number of steps walked daily assessed by actigraphy

CONTACTS AND LOCATIONS:
Locations (1):
- CHu Saint Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No